CLINICAL TRIAL: NCT06492460
Title: A Multicenter, Randomized Controlled, Non-inferior Phase 3 Clinical Trial of 2 Courses of Concurrent Cisplatin Chemoradiotherapy Versus 3 Courses After Surgery for High-risk Head and Neck Squamous Cell Carcinoma
Brief Title: 2 Courses of Concurrent Cisplatin Chemoradiotherapy After Surgery for High-risk Head and Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Hunan Cancer Hospital (Other); Guilin Medical University, China (Other); Jiangsu Cancer Institute & Hospital (Other); Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Lei Chen, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SL-B2024-323-02
Record Dates: First submitted 2024-07-02; First posted 2024-07-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Concurrent chemoradiotherapy; Cisplatin; postoperative head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2 courses of cisplatin chemoradiotherapy arm (Experimental): Patients will receive intensity modulated radiotherapy (total dose: > 66 Gy, split dose: 2-2.2 Gy/ time, once a day, 5 times a week) plus concurrent Cisplatin chemotherapy (100 mg/m2 intravenous injection,once every 3 weeks, twice in total, on days 1 and 22).
  Interventions: Drug: Drug：Cisplatin
- 3 courses of cisplatin chemoradiotherapy arm (Experimental): Patients will receive intensity modulated radiotherapy (total dose: > 66 Gy, split dose: 2-2.2 Gy/ time, once a day, 5 times a week) plus concurrent Cisplatin chemotherapy (100 mg/m2 intravenous injection,once every 3 weeks, once every 3 weeks, 3 times in total, days 1, 22, and 43).
  Interventions: Drug: Drug：Cisplatin

INTERVENTIONS:
Drug: Drug：Cisplatin — Concurrent Cisplatin chemotherapy (100 mg/m2 intravenous injection,once every 3 weeks, twice in total, on days 1 and 22) will be given plus intensity modulated radiotherapy
  Other Names: CDDP Drug

SUMMARY:
The main objective of this trial was to determine the value of 2 courses of cisplatin concurrent chemotherapy in postoperative adjuvant radiotherapy for high-risk head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
The main objective of the trial was to evaluate whether the 3-year failure-free survival (FFS) rate in patients with high-risk head and neck squamous cell carcinoma treated with adjuvant radiotherapy and 2 courses of concurrent cisplatin chemotherapy after surgery was no less than 10% compared with 3 courses of concurrent cisplatin chemotherapy. The secondary objective was to evaluate efficacy and toxicity of 2 courses of concurrent cisplatin chemotherapy (100mg/m2, days 1 and 22) during adjuvant intensity-modulated radiation therapy will be compared with 3 courses of concurrent cisplatin chemotherapy (100mg/m2, days 1, 22 and 43).

ELIGIBILITY:
Inclusion Criteria:

A. The pathological type is head and neck squamous cell carcinoma

* Stages III and IV

B. Radical surgery has been performed with high risk factors (one of below)

* extracapsular invasion of cervical metastatic lymph nodes
* positive incisional margin or inadequate incisional margin safety distance

C. No evidence of distant metastasis (M0).

D. Functional status: Karnofsky scale (KPS) > 70.

E. Normal bone marrow function:

* white blood cell count > 4×109/L
* hemoglobin > 120g/L in males, 110g/L in females
* platelet count > 100×109/L

G. Normal liver function:

* alanine aminotransferase (ALT), aspartate aminotransferase (AST) < 1.5 times the upper limit of normal (ULN)
* alkaline phosphatase (ALP) < 2.5×ULN
* bilirubin < ULN.

H. Normal renal function: creatinine clearance > 60 ml/min.

I. Patients must be informed of the basic contents of this study and sign informed consent.

Exclusion Criteria:

A. Age >70 years or <18 years.

B. Treatment is palliative.

C. Previous chemotherapy (except induction chemotherapy prior to surgery).

D. Previous radiation therapy.

E. Women who are pregnant or breastfeeding

F. Previous history of malignant tumor.

G. With other serious medical conditions that may pose a greater risk or affect compliance with the test. Examples include:

* unstable heart disease that requires treatment
* kidney disease
* chronic hepatitis
* poorly controlled diabetes (fasting blood glucose > 1.5×ULN)
* mental illness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2029-09-20 (Estimated); Study Completion 2033-07-17 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3 years
  calculated from enrolment to the date of locoregional recurrence,distant metastasis,or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  calculated from enrolment to the date of death from any cause.
Distant metastasis-free survival(DMFS) | 3 years
  calculated from enrolment to the date of first distant metastasis.
locoregional recurrence-free survival (LRRFS) | 3 years
  calculated from enrolment to the date of locoregional persistence or 1st locoregional recurrence.
Quality of life (QoL) | 3 years
  The change of QoL from randomization to the start of radiotherapy,the end of radiotherapy,13-16 weeks after radiotherapy,2 years and 3 years after randomization. The EORTC QoL questionnaire-C30(EORTC quality of life questionnaire-C30#version 3.0 will be used. This questionnaire comprises 30 questions,24 of which are aggregated into nine multi- question scales,that is,five functioning scales (e.g.,physical),three symptom scales (e.g.,fatigue)and one global health status scale. The remaining six single-question (e.g.,dyspnoea)scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Chen, M.D, Principal Investigator — Sun Yat-sen University
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Affiliated Hospital of Guilin Medical College, Guilin, Guangxi
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital, Central South University, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Wu C, Li M, Meng H, Liu Y, Niu W, Zhou Y, Zhao R, Duan Y, Zeng Z, Li X, Li G, Xiong W, Zhou M. Analysis of status and countermeasures of cancer incidence and mortality in China. Sci China Life Sci. 2019 May;62(5):640-647. doi: 10.1007/s11427-018-9461-5. Epub 2019 Mar 12. PMID 30900169
- [Background] Bernier J, Domenge C, Ozsahin M, Matuszewska K, Lefebvre JL, Greiner RH, Giralt J, Maingon P, Rolland F, Bolla M, Cognetti F, Bourhis J, Kirkpatrick A, van Glabbeke M; European Organization for Research and Treatment of Cancer Trial 22931. Postoperative irradiation with or without concomitant chemotherapy for locally advanced head and neck cancer. N Engl J Med. 2004 May 6;350(19):1945-52. doi: 10.1056/NEJMoa032641. PMID 15128894
- [Background] Cooper JS, Pajak TF, Forastiere AA, Jacobs J, Campbell BH, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Machtay M, Ensley JF, Chao KS, Schultz CJ, Lee N, Fu KK; Radiation Therapy Oncology Group 9501/Intergroup. Postoperative concurrent radiotherapy and chemotherapy for high-risk squamous-cell carcinoma of the head and neck. N Engl J Med. 2004 May 6;350(19):1937-44. doi: 10.1056/NEJMoa032646. PMID 15128893
- [Background] Bernier J, Cooper JS, Pajak TF, van Glabbeke M, Bourhis J, Forastiere A, Ozsahin EM, Jacobs JR, Jassem J, Ang KK, Lefebvre JL. Defining risk levels in locally advanced head and neck cancers: a comparative analysis of concurrent postoperative radiation plus chemotherapy trials of the EORTC (#22931) and RTOG (# 9501). Head Neck. 2005 Oct;27(10):843-50. doi: 10.1002/hed.20279. PMID 16161069
- [Background] Cooper JS, Zhang Q, Pajak TF, Forastiere AA, Jacobs J, Saxman SB, Kish JA, Kim HE, Cmelak AJ, Rotman M, Lustig R, Ensley JF, Thorstad W, Schultz CJ, Yom SS, Ang KK. Long-term follow-up of the RTOG 9501/intergroup phase III trial: postoperative concurrent radiation therapy and chemotherapy in high-risk squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2012 Dec 1;84(5):1198-205. doi: 10.1016/j.ijrobp.2012.05.008. Epub 2012 Jun 30. PMID 22749632
- [Background] Hartford AC, Palisca MG, Eichler TJ, Beyer DC, Devineni VR, Ibbott GS, Kavanagh B, Kent JS, Rosenthal SA, Schultz CJ, Tripuraneni P, Gaspar LE; American Society for Therapeutic Radiology and Oncology; American College of Radiology. American Society for Therapeutic Radiology and Oncology (ASTRO) and American College of Radiology (ACR) Practice Guidelines for Intensity-Modulated Radiation Therapy (IMRT). Int J Radiat Oncol Biol Phys. 2009 Jan 1;73(1):9-14. doi: 10.1016/j.ijrobp.2008.04.049. No abstract available. PMID 19100920
- [Background] Lee NY, de Arruda FF, Puri DR, Wolden SL, Narayana A, Mechalakos J, Venkatraman ES, Kraus D, Shaha A, Shah JP, Pfister DG, Zelefsky MJ. A comparison of intensity-modulated radiation therapy and concomitant boost radiotherapy in the setting of concurrent chemotherapy for locally advanced oropharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2006 Nov 15;66(4):966-74. doi: 10.1016/j.ijrobp.2006.06.040. PMID 17145527
- [Background] Dogan N, King S, Emami B, Mohideen N, Mirkovic N, Leybovich LB, Sethi A. Assessment of different IMRT boost delivery methods on target coverage and normal-tissue sparing. Int J Radiat Oncol Biol Phys. 2003 Dec 1;57(5):1480-91. doi: 10.1016/s0360-3016(03)01569-4. PMID 14630288
- [Background] Lee NY, O'Meara W, Chan K, Della-Bianca C, Mechalakos JG, Zhung J, Wolden SL, Narayana A, Kraus D, Shah JP, Pfister DG. Concurrent chemotherapy and intensity-modulated radiotherapy for locoregionally advanced laryngeal and hypopharyngeal cancers. Int J Radiat Oncol Biol Phys. 2007 Oct 1;69(2):459-68. doi: 10.1016/j.ijrobp.2007.03.013. Epub 2007 May 9. PMID 17493769
- [Background] Wu Q, Mohan R, Morris M, Lauve A, Schmidt-Ullrich R. Simultaneous integrated boost intensity-modulated radiotherapy for locally advanced head-and-neck squamous cell carcinomas. I: dosimetric results. Int J Radiat Oncol Biol Phys. 2003 Jun 1;56(2):573-85. doi: 10.1016/s0360-3016(02)04617-5. PMID 12738335
- [Background] Adelstein DJ, Moon J, Hanna E, Giri PG, Mills GM, Wolf GT, Urba SG. Docetaxel, cisplatin, and fluorouracil induction chemotherapy followed by accelerated fractionation/concomitant boost radiation and concurrent cisplatin in patients with advanced squamous cell head and neck cancer: A Southwest Oncology Group phase II trial (S0216). Head Neck. 2010 Feb;32(2):221-8. doi: 10.1002/hed.21179. PMID 19557750
- [Background] Lefebvre JL, Pointreau Y, Rolland F, Alfonsi M, Baudoux A, Sire C, de Raucourt D, Malard O, Degardin M, Tuchais C, Blot E, Rives M, Reyt E, Tourani JM, Geoffrois L, Peyrade F, Guichard F, Chevalier D, Babin E, Lang P, Janot F, Calais G, Garaud P, Bardet E. Induction chemotherapy followed by either chemoradiotherapy or bioradiotherapy for larynx preservation: the TREMPLIN randomized phase II study. J Clin Oncol. 2013 Mar 1;31(7):853-9. doi: 10.1200/JCO.2012.42.3988. Epub 2013 Jan 22. PMID 23341517
- [Background] Rades D, Kronemann S, Meyners T, Bohlen G, Tribius S, Kazic N, Schroeder U, Hakim SG, Schild SE, Dunst J. Comparison of four cisplatin-based radiochemotherapy regimens for nonmetastatic stage III/IV squamous cell carcinoma of the head and neck. Int J Radiat Oncol Biol Phys. 2011 Jul 15;80(4):1037-44. doi: 10.1016/j.ijrobp.2010.03.033. Epub 2010 Jul 16. PMID 20638185
- [Background] Lu HJ, Yang CC, Wang LW, Chu PY, Tai SK, Chen MH, Yang MH, Chang PM. Modified weekly cisplatin-based chemotherapy is acceptable in postoperative concurrent chemoradiotherapy for locally advanced head and neck cancer. Biomed Res Int. 2015;2015:307576. doi: 10.1155/2015/307576. Epub 2015 Feb 22. PMID 25793192
- [Background] Geiger JL, Lazim AF, Walsh FJ, Foote RL, Moore EJ, Okuno SH, Olsen KD, Kasperbauer JL, Price DL, Garces YI, Ma DJ, Neben-Wittich MA, Molina JR, Garcia JJ, Price KA. Adjuvant chemoradiation therapy with high-dose versus weekly cisplatin for resected, locally-advanced HPV/p16-positive and negative head and neck squamous cell carcinoma. Oral Oncol. 2014 Apr;50(4):311-8. doi: 10.1016/j.oraloncology.2014.01.001. Epub 2014 Jan 24. PMID 24467937
- [Background] Yau TK, Lee AW, Wong DH, Yeung RM, Chan EW, Ng WT, Tong M, Soong IS. Induction chemotherapy with cisplatin and gemcitabine followed by accelerated radiotherapy and concurrent cisplatin in patients with stage IV(A-B) nasopharyngeal carcinoma. Head Neck. 2006 Oct;28(10):880-7. doi: 10.1002/hed.20421. PMID 16721741
- [Background] Marks LB, Yorke ED, Jackson A, Ten Haken RK, Constine LS, Eisbruch A, Bentzen SM, Nam J, Deasy JO. Use of normal tissue complication probability models in the clinic. Int J Radiat Oncol Biol Phys. 2010 Mar 1;76(3 Suppl):S10-9. doi: 10.1016/j.ijrobp.2009.07.1754. PMID 20171502
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Cox JD, Stetz J, Pajak TF. Toxicity criteria of the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). Int J Radiat Oncol Biol Phys. 1995 Mar 30;31(5):1341-6. doi: 10.1016/0360-3016(95)00060-C. No abstract available. PMID 7713792
- [Background] Bacchetti P, Leung JM. Sample size calculations in clinical research. Anesthesiology. 2002 Oct;97(4):1028-9; author reply 1029-32. doi: 10.1097/00000542-200210000-00050. No abstract available. PMID 12357184